CLINICAL TRIAL: NCT02266810
Title: The PROGRESS Study: Safety and Efficacy of the Propel Mini and Propel Nova Steroid-Eluting Sinus Implants Following Surgical Opening of the Frontal Sinus for Chronic Sinusitis: A Randomized Blinded Controlled Study
Brief Title: Safety and Efficacy of the Propel Mini and Propel Nova Steroid-Eluting Sinus Implant in Frontal Sinus
Acronym: PROGRESS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intersect ENT (Industry)
Collaborators: Advance Research Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P500-0514
Record Dates: First submitted 2014-09-15; First posted 2014-10-17 (Estimated); Results first posted 2017-10-06 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2017-10

CONDITIONS: Chronic Sinusitis

STUDY DESIGN:
Intervention Model Description: Intra-patient control
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- PROPEL Mini Sinus Implant (Experimental): Propel Mini placed in frontal sinus opening following ESS
  Interventions: Device: PROPEL Mini Sinus Implant.
- Sinus Surgery alone: cohort 1 (Active Comparator): Sinus Surgery only: cohort 1: ESS with standard post-operative care.
  Interventions: Procedure: Sinus Surgery alone
- PROPEL Nova Sinus Implant (Experimental): Propel Nova placed in frontal sinus opening following ESS
  Interventions: Device: Propel Nova Sinus Implant
- Sinus Surgery alone: cohort 2 (Active Comparator): Sinus Surgery only: cohort 2: ESS with standard post-operative care.
  Interventions: Procedure: Sinus Surgery alone

INTERVENTIONS:
Device: PROPEL Mini Sinus Implant. — Placement of sinus implant following frontal sinus surgery
  Arms: PROPEL Mini Sinus Implant
Procedure: Sinus Surgery alone — Sinus surgery only, without implant placement
  Arms: Sinus Surgery alone: cohort 1; Sinus Surgery alone: cohort 2
Device: Propel Nova Sinus Implant — Placement of sinus implant following frontal sinus surgery
  Other Names: PROPEL contour Sinus Implant
  Arms: PROPEL Nova Sinus Implant

SUMMARY:
The objective of the PROGRESS Study is to assess the safety and efficacy of the Propel Mini and Propel Nova steroid-eluting Sinus Implants when placed in the frontal sinus opening following frontal sinus surgery in patients with chronic sinusitis.

DETAILED DESCRIPTION:
This is a prospective, randomized, blinded, controlled, multicenter study enrolling two consecutive cohorts of up to 80 patients each (Propel Mini cohort followed by Propel Nova cohort). The study patients will undergo implant placement on one side following ESS that includes bilateral frontal sinus surgery by traditional surgical technique or balloon dilation.

ELIGIBILITY:
Inclusion Criteria:

* Patient has CRS confirmed by CT scan and defined as symptoms lasting longer than 12 consecutive weeks in duration with inflammation of the mucosa of the nose and paranasal sinuses.
* Patient has a clinical indication for and has consented to ESS including bilateral frontal sinus surgery.
* Chronic sinusitis diagnosis confirmed and documented by CT scan within 6 months of the procedure.
* Patient has bilateral disease in both frontal sinuses confirmed by Lund-Mackay score of ≥1 on each side.
* Planned sinus surgery includes bilateral ethmoidectomy (if judged necessary) and frontal sinus enlargement using Draf II (A or B) dissection or balloon dilation, with minimum of 5-mm diameter opening created.
* Technique used for frontal sinus surgery is the same on both sides (e.g. surgical dissection alone bilaterally, balloon dilation alone bilaterally, or both bilaterally)
* Septoplasty for access to the ostio-meatal complex is permitted.
* ESS including bilateral frontal sinus surgery has been successfully completed without significant complication that, in the opinion of the investigator, would confound study results, and the patient's anatomy remains amenable to implant placement.

Exclusion Criteria:

* Known history of immune deficiency such as immunoglobin G or A subclass deficiency, or Human Immunodeficiency Virus (HIV)
* Oral-steroid dependent condition such as chronic obstructive pulmonary disease (COPD) or asthma or other condition
* Known history of allergy or intolerance to corticosteroids or mometasone furoate
* Clinical evidence of acute bacterial sinusitis
* Clinical evidence or suspicion of invasive fungal sinusitis (e.g., bone erosion on CT scan, necrotic sinus tissue)
* Active viral illness
* Concurrent condition requiring active chemotherapy and/or immunotherapy management for the disease
* Clinical evidence of disease or condition expected to compromise survival or ability to complete follow-up assessments during the 90 day follow-up period
* Currently participating in another clinical trial
* History of insulin dependent diabetes mellitus
* Patient has previously undergone ESS and experienced a CSF leak or has compromised vision as a result of a complication in a prior ESS procedure
* Significant complication during the current frontal sinus surgery procedure such as excessive blood loss, CSF leak or punctured lamina papyracea
* Current ESS including frontal sinus surgery is aborted for any reason.
* At least one side is not amenable for implant placement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2014-09; Primary Completion 2016-04 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy L. Smith, MD, MPH, Principal Investigator — Oregon Health and Science University; Amber U. Luong, MD, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (10):
- United States (10):
  - Sacramento Ear, Nose and Throat, Sacramento, California
  - Breathe Clear Institute of Sinus and Allergy Relief, Torrance, California
  - The Connecticut Center for Advanced ENT Care, Norwalk, Connecticut
  - George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - ENT of Georgia, Atlanta, Georgia
  - Advanced ENT and Allergy, Louisville, Kentucky
  - Albany ENT and Allergy, Albany, New York
  - Oregon Health and Science University, Portland, Oregon
  - University of Texas Health Science Center at Houston, Houston, Texas
  - East Virginia Medical School, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Smith TL, Singh A, Luong A, Ow RA, Shotts SD, Sautter NB, Han JK, Stambaugh J, Raman A. Randomized controlled trial of a bioabsorbable steroid-releasing implant in the frontal sinus opening. Laryngoscope. 2016 Dec;126(12):2659-2664. doi: 10.1002/lary.26140. Epub 2016 Jul 1. PMID 27363723
- [Derived] Luong A, Ow RA, Singh A, Weiss RL, Han JK, Gerencer R, Stolovitzky JP, Stambaugh JW, Raman A. Safety and Effectiveness of a Bioabsorbable Steroid-Releasing Implant for the Paranasal Sinus Ostia: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2018 Jan;144(1):28-35. doi: 10.1001/jamaoto.2017.1859. Epub 2017 Nov 2. PMID 29098299

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: sinus sides
Groups:
- PROPEL Mini Sinus Implant: This study will use an intra-patient design. Each patient will undergo placement of one implant. The untreated side will represent the control. The side of placement will be randomly assigned.
  PROPEL Mini Sinus Implant: Placement of sinus implant following frontal sinus surgery
- PROPEL Nova Sinus Implant: This study will use an intra-patient design. Each patient will undergo placement of one implant. The untreated side will represent the control. The side of placement will be randomly assigned.
  PROPEL Nova Sinus Implant: Placement of sinus implant following frontal sinus surgery
Period: Overall Study
Arm/Group | PROPEL Mini Sinus Implant | PROPEL Nova Sinus Implant
Started | 80; 160 sinus sides (sinus sides) | 80; 160 sinus sides (sinus sides)
Completed | 79; 158 sinus sides (sinus sides) | 79; 158 sinus sides (sinus sides)
Not Completed | 1; 2 sinus sides | 1; 2 sinus sides

BASELINE CHARACTERISTICS:
Population: This is an intra-patient design where one sinus side of the patient is randomized to receive the treatment while the contralateral sinus side acts as the control.
Groups:
- PROPEL Mini Sinus Implant and No Implant Cohort 1; PROPEL Nova Sinus Implant and No Implant Cohort 2: This study will use an intra-patient design. Each patient will undergo placement of one implant. The untreated side will represent the control. The side of placement will be randomly assigned.
  PROPEL Mini or Nova Sinus Implant.: Placement of sinus implant following frontal sinus surgery
- Total: Total of all reporting groups
Arm/Group | PROPEL Mini Sinus Implant and No Implant Cohort 1 | PROPEL Nova Sinus Implant and No Implant Cohort 2 | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (13.91) | 49.5 (13.36) | 49.7 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 27 | 61
  Male | 46 | 53 | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 80 | 77 | 157
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 9 | 21
  White | 62 | 68 | 130
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 80 | 80 | 160

OUTCOME MEASURES:

1. Primary Outcome: Percent of Sinuses That Require Post-operative Interventions (Propel Mini Cohort)
Description: The reduction in need for post-operative interventions at Day 30, as determined by an independent blinded sinus surgeon based on video-endoscopy reviews.
  Need for Post-Operative Intervention is a composite endpoint that includes: surgical intervention required to debride obstructive adhesions or scar tissue formation in the Frontal sinus opening(defined as grade 2 or 3 on the adhesion/scarring scale), and/or oral steroid intervention warranted to resolve recurrent inflammation and polypoid edema in the frontal recess/FSO (Yes/No response).
Time Frame: Day 30
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percent sinuses requiring intervention
Groups:
- Sinus Surgery Only: Cohort 1: Sinus surgery with standard post-operative care.
  Sinus Surgery alone: Sinus surgery only, without implant placement
Arm/Group | PROPEL Mini Sinus Implant | Sinus Surgery Only: Cohort 1
Number analyzed (Participants) | 67 | 67
percent sinuses requiring intervention | 38.8 [27.1 to 51.5] | 62.7 [50.0 to 74.2]

2. Primary Outcome: Percent of Sinuses That Require Post-operative Interventions (Propel Nova Cohort)
Description: as for outcome 1
Time Frame: Day 30
Population: Of the 80 patients who had their endoscopy recorded at day 30 for grading by independent reviewer; 19 patients could not be included in the test due to missing data. Data were considered missing if the independent reviewer could not grade a video on one or both treatment sinus sides.
Measure: Number (95% Confidence Interval); unit: percentage sinus requiring intervention
Groups:
- Sinus Surgery Only: Cohort 2: Sinus surgery with standard post-operative care.
  Sinus Surgery alone: Sinus surgery only, without implant placement
Arm/Group | PROPEL Nova Sinus Implant | Sinus Surgery Only: Cohort 2
Number analyzed (Participants) | 61 | 61
percentage sinus requiring intervention | 11.5 [4.7 to 22.2] | 32.8 [21.3 to 46.0]

3. Secondary Outcome: Need for Post-operative Interventions (Propel Mini Cohort)
Description: Need for post-operative interventions by clinical investigators at Day 30
  Need for Post-Operative Intervention is a composite endpoint that includes: surgical intervention required to debride obstructive adhesions or scar tissue formation in the FSO (defined as grade 2 or 3 on the adhesion/scarring scale), and/or oral steroid intervention warranted to resolve recurrent inflammation and polypoid edema in the frontal recess/FSO (Yes/No response).
Time Frame: Day 30
Measure: Number (95% Confidence Interval); unit: percentage of evaluable sinuses
Units Other Than Participants: sinus sides
Groups:
- Sinus Surgery Only: Cohort 1: This study will use an intra-patient design. Each patient will undergo placement of one implant. The untreated side will represent the control. The side of placement will be randomly assigned.
  Sinus Surgery only: Sinus surgery only, without implant placement
Arm/Group | PROPEL Mini Sinus Implant | Sinus Surgery Only: Cohort 1
Number analyzed (Participants) | 80 | 80
Number analyzed (sinus sides) | 79 | 79
percentage of evaluable sinuses | 16.5 [9.1 to 26.5] | 41.8 [30.8 to 53.4]

4. Secondary Outcome: Need for Surgical Interventions (Propel Mini Cohort)
Description: Need for Surgical Interventions by clinical investigators at Day 30.
  Need for surgical interventions was prospectively defined as Adhesion/scarring grades of 2 and 3.
  Adhesions/Scarring was assessed based on a 4-point scale as follows:
  0= No visible granulation/scarring in the FSO
  1. Minimal amount of granulation, scarring or contraction observed but not obstructing the FSO (intervention not warranted)
  2. Moderate amount of obstructive granulation, scarring or contraction present in the FSO (intervention is warranted)
  3. Significant amount of scarring or contraction causing obstruction of the FSO requiring intervention (likely to compromise patency if not removed)
Time Frame: Day 30
Measure: Number; unit: percentage of evaluable sinuses
Units Other Than Participants: sinus sides
Arm/Group | PROPEL Mini Sinus Implant | Sinus Surgery Only: Cohort 1
Number analyzed (Participants) | 80 | 80
Number analyzed (sinus sides) | 75 | 75
percentage of evaluable sinuses | 4.0 | 16.0

5. Secondary Outcome: Inflammation (Propel Mini Cohort)
Description: The degree of inflammation present in the frontal recess/FSO was evaluated by clinical investigators using a 100-mm VAS ranging from 0 defined as no visible inflammation to 100 defined as severe inflammation, involving extensive erythema, edema, or polyposis.
Time Frame: Day 30
Measure: Mean (Standard Deviation); unit: 100-mm VAS
Units Other Than Participants: sinus sides
Arm/Group | PROPEL Mini Sinus Implant | Sinus Surgery Alone: Cohort 1
Number analyzed (Participants) | 80 | 80
Number analyzed (sinus sides) | 79 | 79
100-mm VAS | 24.7 (27.02) | 41.3 (29.34)

6. Secondary Outcome: Occlusion/Restenosis (Propel Mini Cohort)
Description: Patency of the FSO was assessed by clinical investigators endoscopically on a 3-point grading scale as follows:
  0=Patent
  1. Restenosed/Partially Occluded
  2. Occluded
Time Frame: Day 30
Measure: Number (95% Confidence Interval); unit: percentage of evaluable sinuses
Units Other Than Participants: sinus sides
Arm/Group | PROPEL Mini Sinus Implant | Sinus Surgery Only: Cohort 1
Number analyzed (Participants) | 80 | 80
Number analyzed (sinus sides) | 76 | 76
percentage of evaluable sinuses | 21.1 [12.5 to 31.9] | 46.1 [34.5 to 57.9]

7. Secondary Outcome: Need for Post-operative Interventions (Propel Nova Cohort)
Description: Need for post-operative interventions by clinical investigators at Day 30.
  Need for Post-Operative Intervention is a composite endpoint that includes: surgical intervention required to debride obstructive adhesions or scar tissue formation in the FSO (defined as grade 2 or 3 on the adhesion/scarring scale by investigators), and/or oral steroid intervention warranted to resolve recurrent inflammation and polypoid edema in the frontal recess/FSO (Yes/No response).
Time Frame: Day 30
Measure: Number (95% Confidence Interval); unit: percentage of evaluable sinuses
Units Other Than Participants: sinus sides
Groups:
- Sinus Surgery Only: Cohort 2: This study will use an intra-patient design. Each patient will undergo placement of one implant. The untreated side will represent the control. The side of placement will be randomly assigned.
  Sinus Surgery only: Sinus surgery only, without implant placement
Arm/Group | PROPEL Nova Sinus Implant | Sinus Surgery Only: Cohort 2
Number analyzed (Participants) | 80 | 80
Number analyzed (sinus sides) | 75 | 75
percentage of evaluable sinuses | 16.0 [8.6 to 26.3] | 33.3 [22.9 to 45.2]

8. Secondary Outcome: Need for Surgical Interventions (Propel Nova Cohort)
Description: Need for Surgical Interventions by clinical investigators at Day 30
  Need for Surgical Interventions by clinical investigators at Day 30.
  Need for surgical interventions was prospectively defined as Adhesion/scarring grades of 2 and 3.
  Adhesions/Scarring was assessed based on a 4-point scale as follows:
  0= No visible granulation/scarring in the FSO
  1. Minimal amount of granulation, scarring or contraction observed but not obstructing the FSO (intervention not warranted)
  2. Moderate amount of obstructive granulation, scarring or contraction present in the FSO (intervention is warranted)
  3. Significant amount of scarring or contraction causing obstruction of the FSO requiring intervention (likely to compromise patency if not removed)
Time Frame: Day 30
Measure: Number; unit: percentage of evaluable sinuses
Units Other Than Participants: sinus sides
Groups:
- PROPEL Nova Sinus Implant: Propel Nova placed in frontal sinus opening following ESS
  PROPEL Nova Sinus Implant.: Placement of sinus implant following frontal sinus surgery
Arm/Group | PROPEL Nova Sinus Implant | Sinus Surgery Only: Cohort 2
Number analyzed (Participants) | 80 | 80
Number analyzed (sinus sides) | 75 | 75
percentage of evaluable sinuses | 4.0 | 14.7

9. Secondary Outcome: Inflammation (Propel Nova Cohort)
Description: as for outcome 5
Time Frame: Day 30
Measure: Mean (Standard Deviation); unit: 100-mm VAS
Units Other Than Participants: sinus sides
Arm/Group | PROPEL Nova Sinus Implant | Sinus Surgery Alone: Cohort 2
Number analyzed (Participants) | 80 | 80
Number analyzed (sinus sides) | 79 | 77
100-mm VAS | 23.1 (24.23) | 35.6 (31.12)

10. Secondary Outcome: Occlusion/Restenosis (Propel Nova Cohort)
Description: as for outcome 6
Time Frame: Day 30
Measure: Number (95% Confidence Interval); unit: percentage of evaluable sinuses
Units Other Than Participants: sinus sides
Arm/Group | PROPEL Nova Sinus Implant | Sinus Surgery Only: Cohort 2
Number analyzed (Participants) | 80 | 80
Number analyzed (sinus sides) | 75 | 75
percentage of evaluable sinuses | 13.3 [6.6 to 23.2] | 36.0 [25.2 to 47.9]

ADVERSE EVENTS:
Time Frame: Propel Mini cohort: 90 days
Arm/Group | PROPEL Mini Sinus Implant | PROPEL Nova Sinus Implant
Serious Adverse Events (participants affected / at risk) | 3/80 | 1/80
Other Adverse Events (participants affected / at risk) | 43/80 | 36/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PROPEL Mini Sinus Implant (N=80) | PROPEL Nova Sinus Implant (N=80)
Cerebrovascular Accident (Vascular disorders) | 0 (0) | 1 (1) — not device-related
Diverticulitis (Infections and infestations) | 1 (1) | 0 — not device related
Respiratory tract infection fungal (Infections and infestations) | 1 (1) | 0 — not device related
deep vein thrombosis (Vascular disorders) | 1 (2) | 0 — not device related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PROPEL Mini Sinus Implant (N=80) | PROPEL Nova Sinus Implant (N=80)
acute sinusitis (Infections and infestations) | 12 (12) | 16 (16) — not device related
chronic sinusitis (Infections and infestations) | 9 (9) | 4 (4) — not device related
upper respiratory tract infection (Infections and infestations) | 5 (5) | 4 (4) — not device related
headache (Nervous system disorders) | 9 (9) | 5 (5) — not device related
presyncope (Nervous system disorders) | 4 (4) | 0 — not device related
epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) — not device related
asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less